CLINICAL TRIAL: NCT03060356
Title: Clinical Trial of Autologous cMET Redirected T Cells Administered Intravenously in Patients With Melanoma & Breast Carcinoma
Brief Title: Autologous T Cells Expressing MET scFv CAR (RNA CART-cMET)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Halt in funding
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 11916, 825376
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Malignant Melanoma; Breast Cancer
MeSH Terms: conditions — Melanoma; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melanoma (Active Comparator): Intravenous infusion 1x10^8 total T cells modified with RNA anti-cMET CAR
  Interventions: Biological: T cells modified with RNA anti -cMET CAR
- Breast (Active Comparator): Intravenous infusion 1x10^8 total T cells modified with RNA anti-cMET CAR
  Interventions: Biological: T cells modified with RNA anti -cMET CAR

INTERVENTIONS:
Biological: T cells modified with RNA anti -cMET CAR — Intravenously administered, RNA electroporated autologous T cells expressing MET chimeric antigen receptors with tandem TCRζ and 4-1BB (TCRζ /4-1BB) co-stimulatory domains

SUMMARY:
This is a pilot study to evaluate feasibility, safety, and preliminary evidence of efficacy for intravenously administered, RNA electroporated autologous T cells expressing MET chimeric antigen receptors with tandem TCRζ and 4-1BB (TCRζ /4-1BB) co-stimulatory domains (referred to as "RNA CART-cMET") in patients with advanced melanoma or breast carcinoma.

DETAILED DESCRIPTION:
This is a pilot study to evaluate feasibility, safety, and preliminary evidence of efficacy for intravenously administered, RNA electroporated autologous T cells expressing MET chimeric antigen receptors with tandem TCRζ and 4-1BB (TCRζ /4-1BB) co-stimulatory domains (referred to as "RNA CART-cMET") in patients with advanced melanoma or breast carcinoma. Subjects will be treated with IV administration of the RNA transduced anti-cMET CAR T cells for a total of up to six doses over a 2 week period.

Each dose is 1x108 total T cells modified with RNA anti-cMET CAR. All subjects in both the melanoma and breast carcinoma arms will receive up to 6 doses of RNA CART-cMET cells, with no lymphodepleting chemotherapy administered prior to cell infusion Cell numbers are based on total cells with a portion of them having CAR expression depending on transduction efficiency and determined by flow cytometry Based on the product release criteria, at least 20% of the total cells will express the anti-cMET CAR. Treatment limiting toxicity (TLT). Adverse event reporting will begin at the start of the first dose of RNA CART-cMET and will continue until 4 months after the first infusion, or until another alternative therapy is initiated, whichever occurs earlier. Subjects will be continually reassessed for evidence of acute and cumulative toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable histologically confirmed stage III/IV melanoma or metastatic or locally advanced unresectable ER and PR negative, HER2 neu nonamplified by IHC and/or FISH breast carcinoma
* cMET expression in ≥ 30% tumor cells as demonstrated on immunohistochemistry analysis at the University of Pennsylvania. MET IHC may be performed on tissue from screening biopsy, or archival slides of a metastatic deposit or primary tumor. Punch biopsy or percutaneous core biopsy will be offered to obtain tissue as required for this purpose.
* Patients must have measureable disease as defined by RECIST 1.1 criteria; must have CT scan of chest, abdomen, pelvis within 1 month of enrollment that demonstrates measurable disease by RECIST 1.1 criteria in a tumor other than the one being potentially biopsied and resected for correlative studies
* Failure of at least one prior standard of care therapy for advanced stage disease
* If previously treated with any form of immunotherapy (including agents targeting PD1 or CTLA4, oncolytic viruses) the last administered treatment must be at least 2 weeks prior to enrollment
* Males or female patients age > 18 years old
* Eastern Cooperative Oncology Group (ECOG) Clinical Performance Status 0 or 1
* Adequate hematologic and organ function as defined by:
* WBC > 3.0 and ANC >1500
* Plt > 75,000 (no transfusion permitted within 2 weeks to achieve this goal)
* Hgb > 9 g/dl (transfusions are permitted to achieve this goal)
* serum creatinine ≤ 1.5 times upper limit of normal
* Total bilirubin ≤ 2times upper limit of normal
* ALT and AST ≤ 2 times upper limit of normal
* Cardiac ejection fraction of >40% as measured by resting echocardiogram
* Women of child bearing potential must have a negative serum or urine pregnancy test and agree to use appropriate contraception from enrollment through the duration of the trial. Men must agree to use appropriate contraception from enrollment through the duration of the trial.
* Patients must provide written informed consent.

Exclusion Criteria:

* Known metastatic tumor encasing a great vessel or at risk for imminently causing spinal cord compression
* Known HIV-1/HIV-2 infection
* Known active infection with Hepatitis B virus or Hepatitis C virus
* Received an experimental therapy within 30 days of enrollment
* Pregnant women or lactating women
* History of alcohol abuse or illicit drug use within 12 months of enrollment
* Clinically significant comorbid disease or other underlying condition, including significant active infection, in the opinion of the PI or sub-investigators, would contraindicate study therapy or interfere with interpretation of study results
* Significant psychiatric disorder and/or any other reason in the Investigator's opinion that would jeopardize protocol compliance or compromise the patient's ability to give informed consent.
* Patients with known allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
* Patients with clinically apparent arrhythmia, or arrhythmias that are not stable on medical management within 2 weeks of the Screening/Enrollment visit.
* Having received prior genetically manipulated T-cells in prior clinical trial
* History of autoimmune disease (including but not limited to: systemic lupus erythematosis, Sjogren syndrome, rheumatoid arthritis, psoriasis multiple sclerosis, inflammatory bowel disease etc).
* History of immune related adverse event with previous immunotherapy.
* Chronic use of therapeutic anti-coagulants such as coumadin, heparin, or lovenox
* Symptomatic or untreated CNS metastases. Pts with previously treated CNS metastases are eligible if lesions are radiographically/clinically stable without requirement of steroids within 4 weeks prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 in melanoma and breast cancer subjects | from day 0 - month 4

SECONDARY OUTCOMES:
Objective overall response rate by clinical exam for visible cutaneous tumors | day 25 and month 4
Objective overall response rate by radiologic imaging using RECIST 1.1 | day 25 and month 4
Estimate the activity of RNA CART-cMET in subjects who receive at least 1 dose of cells by objective response rate using RECIST 1.1 criteria | day -7 and day 11
Estimate the activity of RNA CART-cMET in subjects who receive at least 1 dose of cells by objective response rate using pathological evaluation of resected or biopsied tissue | day -7 and day 11

CONTACTS AND LOCATIONS:
Overall Officials: Tara C. Mitchell, MD, Principal Investigator — University of Pennaylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shah PD, Huang AC, Xu X, Orlowski R, Amaravadi RK, Schuchter LM, Zhang P, Tchou J, Matlawski T, Cervini A, Shea J, Gilmore J, Lledo L, Dengel K, Marshall A, Wherry EJ, Linette GP, Brennan A, Gonzalez V, Kulikovskaya I, Lacey SF, Plesa G, June CH, Vonderheide RH, Mitchell TC. Phase I Trial of Autologous RNA-electroporated cMET-directed CAR T Cells Administered Intravenously in Patients with Melanoma and Breast Carcinoma. Cancer Res Commun. 2023 May 9;3(5):821-829. doi: 10.1158/2767-9764.CRC-22-0486. eCollection 2023 May. PMID 37377890